CLINICAL TRIAL: NCT04899271
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of 400 mg Twice a Day Oral Ladarixin in Patients With New-onset Type 1 Diabetes and Preserved Beta-cell Function at Baseline.
Brief Title: A Study to Assess Efficacy/Safety of Ladarixin in Type 1 Diabetes Patients With Preserved ß-cell Function at Baseline.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDX0419; 2020-002966-15 (EudraCT Number)
Record Dates: First submitted 2021-05-10; First posted 2021-05-24 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: New-onset Type 1 Diabetes
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Appearance, including packaging and labelling, of the IMP (capsules, packaging) will not allow to recognize actual treatment (either ladarixin or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ladarixin (Experimental): The treatment group received 400 mg b.i.d. for 13 cycles of 14 days on/14 days off)
  Interventions: Drug: Ladarixin
- Placebo (Placebo Comparator): The control group received matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ladarixin — 400 mg b.i.d. for 13 cycles of 14 days on/14 days off
  Other Names: LDX
  Arms: Ladarixin
Other: Placebo — Placebo was administered orally with the same scheme of administration of LDX to preserve blinding
  Arms: Placebo

SUMMARY:
The objective of this clinical trial was to assess whether ladarixin treatment is effective to improve glycemic control in newly diagnosed Type 1 Diabetes (T1D) adult patients with preserved β-cell function.

The safety of ladarixin in the specific clinical setting was also evaluated.

DETAILED DESCRIPTION:
This was a phase II clinical trial designed as a randomized, double-blind, placebo-controlled, multicenter study to evaluate whether ladarixin is effective in preserving β-cell function and slowing-down the progression of T1D in adult patients with new-onset T1D and preserved β- cell function (fasting C-peptide ≥0.205 nmol/L) at baseline.

Seventy-five (75) patients were to be randomized based on an unbalanced randomization allocation ratio (2:1) to ladarixin hard gelatine capsules for oral administration (2 x 200 mg two times a day [b.i.d.] for 13 cycles of 14 days on/14 days off) or matched placebo. Assuming a 10% drop-out rate, approximately 84 patients were expected to be enrolled and to be treated for 1 year.

Each patient was to be involved in the study for a run-in period (screening and baseline assessments) followed by a randomization visit, a treatment period of 12 months, and a post-randomization period up to 18 months from the 1st treatment dose.

The study enrolment was stopped, though, on 28 March 2022, due to low enrolment rate, at the randomization of the 25th patient. The study terminated early, on 11 October 2023 (LPLV).

Due to the early termination of the study, efficacy analyses were reduced in scope given the limited sample size of the study compared with the one expected.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-45 years, inclusive;
2. New-onset T1D (1st IMP dose within 100 days from 1st insulin administration);
3. Positive for at least one diabetes-related auto-antibody (anti-GAD; IAA, if obtained within 10 days of the onset of insulin therapy; IA-2 antibody; ZnT8);
4. Require, or has required at some time, insulin therapy through multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII);
5. Fasting C peptide ≥0.205nmol/L on two occasions;
6. Patient able to comply with all protocol procedures for the duration of the study, including scheduled follow-up visits and examinations;
7. Patients who have given written informed consent prior of any study-related procedure not part of standard medical care.

Exclusion Criteria:

1. Any other chronic disease, including type 2 diabetes, apart from autoimmune hypothyroidism requiring thyroid hormone replacement only; patients with severe (myxedema) disease potentially requiring immunosuppressive therapy will be excluded;
2. Moderate to severe renal impairment as per estimated Glomerular Filtration Rate (eGFR) 60 mL/min/1.73 m2, as determined using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation (see Appendix 14.4.3);
3. Hepatic dysfunction defined by increased ALT/AST > 3 x upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L];
4. Hypoalbuminemia defined as serum albumin < 3 g/dL;
5. QTcF > 470 msec;
6. A history of significant cardiovascular disease/abnormality
7. Occurrence of an episode of ketoacidosis or hypoglycemic coma in the past 2 weeks;
8. Known hypersensitivity to non-steroidal anti-inflammatory drugs;
9. Concomitant treatment with drugs metabolized by CYP2C9 with a narrow therapeutic index [i.e., phenytoin, warfarin, sulphanylurea hypoglycemics (e.g. tolbutamide, glipizide, glibenclamide/glyburide, glimepiride, nateglinide) and high dose of amitriptyline (>50 mg/day)];
10. Previous (within 2 weeks prior to randomization) and concomitant treatment with antidiabetic agents as metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors, SGLT2-inhibitors or amylin, or any medications known to influence glucose tolerance (e.g. beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine antimalarial drugs, lithium, niacin, etc.);
11. Past (within 1 month prior to randomization) or current administration of any immunosuppressive medications (including oral, inhaled or systemically injected steroids) and use of any investigational agents, including any agents that impact the immune response or the cytokine system;
12. Significant systemic infection during the 4 weeks before the first dose of the study drug (e.g., infection requiring hospitalization, major surgery, or IV antibiotics to resolve; other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion);
13. Hepatitis A (IgM), hepatitis B (not due to immunization), hepatitis C and HIV positive serologic status Serologic evidence of current infectious liver disease (hepatitis A, B, or C), including anti hepatitis A virus (immunoglobulin M), hepatitis B surface antigen, or anti hepatitis C virus and HIV;
14. Pregnant or breast feeding women. Unwillingness to use effective contraceptive measures up to 2 months after the end of study drug administration (females and males). Effective contraceptive measures include a hormonal birth control (e.g. oral pills, long term injections, vaginal ring, patch); the intrauterine device (IUD); a double barrier method (e.g. condom or diaphragm plus spermicide foam).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Minnella, MD, Study Director — Dompé Farmaceutici
Locations (16):
- United States (2):
  - University of Colorado School of Medicine - Barbara Davis Center for Childhood Diabetes (BDC) - Specialty Clinic, Aurora, Colorado
  - Atlanta Diabetes Associates (ADA), Atlanta, Georgia
- Universitair Ziekenhuis Brussel (UZB), Jette, Belgium
- Georgia (2):
  - National Center for Diabetes Research LTD, Tbilisi
  - National Institute of Endocrinology LTD, Tbilisi
- Germany (3):
  - Universitaetsklinikum Gessen und Marburg GmbH - Medizinische Klinik und Poliklinik III, Glessen
  - St. Josefskrankenhaus Diabestesinstitut Heidelberg, Heidelberg
  - Institut fuer Diabetes forschung in Muenster (IDFM), Münster
- Italy (6):
  - Azienda Ospedaliero-Universitaria Conzorziale Policlinico di Bari, Bari
  - Università degli Studi Magna Graecia di Catanzaro, Azienda Ospedaliero-Universitaria Mater Domini, Catanzaro
  - Universitá degli Studi di Milano - Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
  - Università Campus Bio-Medico di Roma (UCBM), Roma
  - "Sapienza" Università di Roma- Azienda Ospedaliero Universitaria Policlinico Umberto I, Rome
- Serbia (2):
  - University of Serbia, Clinic for Endocrinology, Diabetes and Metabolic Diseases, Belgrade
  - University of Kragujevac, Clinic for internal diseases, Center for endocrinology, diabetes and metabolic diseases, Kragujevac

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of patients randomized and treated was lower than planned in the study protocol. The Sponsor decided to stop patient enrolment on 28 March 2022, due to the recruitment rate being lower than expected. At the time of recruitment closure, 25 patients had been randomized compared with the 75 planned.
Pre-assignment Details: Overall, 80 participants were screened, having signed the informed consent form. Out of these, 52 participants (65.0%) did not meet eligibility criteria (screen failure) and 3 participants (3.8%) withdrew their consent, making a total of 55 participants (68.8%) not enrolled and thus not randomized.
Groups:
- Ladarixin: The treatment group will receive 400 mg b.i.d. for 13 cycles of 14 days on/14 days off)
  Ladarixin: 400 mg b.i.d. for 13 cycles of 14 days on/14 days off
- Placebo: The control group will receive matched placebo
  Placebo: Placebo will be administered orally with the same scheme of administration of LDX to preserve blinding
Period: Overall Study
Arm/Group | Ladarixin | Placebo
Started | 18 | 7
Received IMP | 18 | 7
FAS Population | 18 | 7
SAF Population | 18 | 7
Completed Week 11 Visit (End of Cycle 3), | 17 | 7
Completed Week 23 Visit (End of Cycle 6) | 16 | 7
Completed Month 6 Visit, | 16 | 7
Completed Week 35 Visit (End of Cycle 9) | 15 | 7
Completed Month 12 Visit (End of Cycle 13), | 15 | 7
Completed (Completed the study (Month 18 visit),) | 15 | 7
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject request/consent withdrawal | 2 | 0

BASELINE CHARACTERISTICS:
Population: FAS population: Full Analysis Set: it consisted of all randomized patients who received at least 1 dose of the IMP (either ladarixin or placebo). The FAS was analyzed according to the Intention To Treat (ITT) principle, i.e., by treatment allocation regardless happening of intercurrent events (treatment policy strategy). The FAS was used for the primary analyses of the study and to present results on efficacy data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ladarixin | Placebo | Total
Number analyzed (Participants) | 18 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 7 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (7.6) | 27.3 (7.7) | 26.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 12 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 7 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
  Italy | 8 | 3 | 11
  Serbia | 5 | 1 | 6
  Germany | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With HbA1c <7% and Daily Insulin Requirement <0.50 IU/Kg/Day at Month 12
Description: The sample size of the study is calculated on the "proportion of patients with a HbA1c < 7% and daily insulin requirement <0.50 IU/Kg/day", a post-hoc composite endpoint derived from data of the phase 2 trial (MEX0114), considering a larger effect size expected from the longer treatment length (one year versus 3 months).
  The time frame for the primary endpoint has been set at Month 12 (Week 52) in order to evaluate the potential of ladarixin effects on a long-term projection.
  Please note that "proportion" is expressed as "count" (number + % of participants)
Time Frame: Month 12 (52±2 weeks)
Population: FAS: The Full Analysis Set consisted of all randomized patients who received at least one dose of the IMP (either ladarixin or placebo). The FAS was analyzed according to the ITT principle, i.e., by treatment allocation regardless happening of intercurrent events (treatment policy strategy). The FAS was used for the primary analyses of the study and to present results on efficacy data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 18 | 7
Participants | 11 | 5
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Test type: Superiority; p = 0.807, Chi-squared

2. Secondary Outcome: Number of Patients With HbA1c < 7% and Daily Insulin Requirement <0.50 IU/Kg/Day at Months 6 and 18
Description: The sample size of the study is calculated on the "proportion of patients with a HbA1c < 7% and daily insulin requirement <0.50 IU/Kg/day", a post-hoc composite endpoint derived from data of the phase 2 trial (MEX0114), considering a larger effect size expected from the longer treatment length (one year versus 3 months). Follow-up is extended up to 18 months to evaluate the potential persistency of any glycemic benefit. Please note that "proportion" is expressed as "count" (number + % of participants)
Time Frame: Month 6 (26±2 weeks) and Month 18 (78±2 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 18 | 7
Participants
  Month 6 | 12 | 6
  Month 18 | 8 | 5
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6; Test type: Superiority; p = 0.746, Chi-squared
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 18; Test type: Superiority; p = 0.201, Chi-squared

3. Secondary Outcome: Number of Patients With a Reduction in HbA1c% > 0.5% From Baseline and Daily Insulin Requirement <0.50 IU/Kg/Day at Months 6, 12 and 18
Description: The number of patients with a reduction in HbA1c% > 0.5% from baseline and daily insulin requirement <0.50 IU/Kg/day was calculated at the hereunder specified timepoints.
Time Frame: Months 6 (26±2 weeks), 12 (52±2 weeks) and 18 (78±2 weeks )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 18 | 7
Participants
  Month 6 | 8 | 4
  Month 12 | 8 | 3
  Month 18 | 6 | 2
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6; Test type: Superiority; p = 0.867, Chi-squared
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 12; Test type: Superiority; p = 0.769, Chi-squared
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Comparison at month 18; Test type: Superiority; p = 0.776, Chi-squared

4. Secondary Outcome: Change From Baseline in 2-hour AUC of C-peptide Response to the MMTT at Months 6, 12 and 18
Description: C-peptide level is a widely used measure of pancreatic beta-cell function and the MMTT is one of the methods for its estimation. AUC stands for Area Under the Curve.
  AUC calculation was based on actual rather scheduled timings and it was calculated using the trapezoidal rule. C-peptide 0-120 min AUC (nmol/L) values were calculated based on all Basal-120min C-peptide values. Unscheduled assessments were excluded from the analysis.
Time Frame: Months 6 (26±2 weeks), 12 (52±2 weeks) and 18 (78±2 weeks)
Population: FAS (Full Analysis Set): all randomized patients who received at least one dose of the IMP (either ladarixin or placebo), analyzed according to the ITT principle. Discrepancies between Overall Number of Participants Analyzed and Number Analyzed for Ladarixin group due to: at Month 6: 2 participants withdrew their consent; at Month 12: 1 additional participant was lost at follow-up (who remained lost at follow-up even for Month 18 visit).
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 16 | 7
nmol/L
  Month 6 | -7.17 (19.33) | -12.70 (16.87)
  Month 12: number analyzed (Participants) | 15 | 7
  Month 12 | 0.25 (23.77) | -0.88 (53.61)
  Month 18: number analyzed (Participants) | 15 | 7
  Month 18 | -2.07 (20.79) | -5.41 (32.52)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6 for change from baseline; Test type: Superiority; p = 0.521, t-test, 2 sided — Assumption of normality was confirmed by Kolmogorov-Smirnov test; the comparison between treatment arms was performed by means of two-sample t-test
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 12 for change from baseline; Test type: Superiority; p = 0.959, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Comparison at month 18 for change from baseline; Test type: Superiority; p = 0.773, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Changes From Baseline in Percentage Glycated Hemoglobin (HbA1c) Levels at Months 6, 12 and 18
Description: HbA1c measurement can be used as a diagnostic test for diabetes providing that stringent quality assurance tests are in place and assays are standardised to criteria aligned to the international reference values, and there are no conditions present which preclude its accurate measurement.
  An HbA1c of 6.5% is recommended as the cut point for diagnosing diabetes. A value of less than 6.5% does not exclude diabetes diagnosed using glucose tests. An A1C test measures the percentage of red blood cells that have glucose-coated hemoglobin.
Time Frame: Months 6 (26±2 weeks), 12 (52±2 weeks) and 18 (78±2 weeks)
Population: FAS (Full Analysis Set): all randomized patients who received at least one dose of the IMP (either ladarixin or placebo), analyzed according to the ITT principle. Discrepancies between Overall Number of Participants Analyzed and Number Analyzed in both arms are due to participants withdrawing consent or with blood samples not collected at timepoints or lost at follow-up.
Measure: Mean (Standard Deviation); unit: percentage HbA1c
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 15 | 7
percentage HbA1c
  Month 6 | -0.67 (0.88) | -0.84 (1.11)
  Month 12: number analyzed (Participants) | 14 | 6
  Month 12 | -0.51 (1.24) | -0.77 (1.28)
  Month 18: number analyzed (Participants) | 15 | 6
  Month 18 | -0.30 (1.55) | -0.33 (0.67)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6 for change from baseline; Test type: Superiority; p = 0.691, t-test, 2 sided; Assumption of normality is confirmed by Kolmogorov-Smirnov test; comparison between treatment arms is performed by means of two-sample t-test
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 12 for change from baseline; Test type: Superiority; p = 0.685, t-test, 2 sided — Assumption of normality is confirmed by Kolmogorov-Smirnov test; comparison between treatment arms is performed by means of two-sample t-test
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Comparison at month 18 for change from baseline; Test type: Superiority; p = 0.640, Wilcoxon (Mann-Whitney) — Assumption of normality is not confirmed by Kolmogorov-Smirnov test; comparison between treatment arms is performed by means of two-sample Mann-Whitney U test

6. Secondary Outcome: Number of Patients With HbA1c < 7% Who Did Not Experience Severe Hypoglycemic Events During Treatment at Months 6,12 and 18
Description: For the purpose of this study, a severe hypoglycaemic event is defined as an event with one of the following symptoms: memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL (3.0 mmol/L) or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: Months 6 (26±2 weeks), 12 (52±2 weeks) and 18 (78±2 weeks)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 15 | 7
Participants
  Month 6 | 7 | 3
  Month 12: number analyzed (Participants) | 14 | 6
  Month 12 | 8 | 3
  Month 18: number analyzed (Participants) | 15 | 6
  Month 18 | 7 | 2
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6; Test type: Superiority; p = 0.867, Chi-squared — Comparison between treatment arms is performed by means of a Chi-squared test
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 12; Test type: Superiority; p = 0.769, Chi-squared — Comparison between treatment arms is performed by means of a Chi-squared test; Comparison between treatment arms is performed by means of a Chi-squared and Fisher's Exact test separated with a /
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Comparison at month 18; Test type: Superiority; p = 0.577, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared test

7. Secondary Outcome: Overall Number of Self-reported Episodes of Severe Hypoglycemia
Description: For the purpose of this study, a severe hypoglycaemic event is defined as an event with one of the following symptoms: memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL (3.0 mmol/L) or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration. Data reported refer to the overall number of episodes recorded by all analyzed patients in the two arms/groups (Ladarixin and placebo).
Time Frame: From baseline to study termination (month 18, week 78)
Population: FAS: The Full Analysis Set consisted of all randomized patients who received at least one dose of the IMP. The FAS was analyzed according to the ITT principle, i.e., by treatment allocation regardless happening of intercurrent events (treatment policy strategy). The FAS was used for the primary analyses of the study and to present results on efficacy data.
Measure: Number; unit: total number of severe hypoglyc episodes
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 18 | 7
total number of severe hypoglyc episodes | 28 | 8
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Test type: Superiority — The effect of treatment on the cumulative number of severe hypoglycemic events was evaluated by means of a Cox proportional hazards model. The Andersen-Gill intensity model with model-based variance was utilized; p = 0.554, Cox proportional hazards model; Analysis is based on Cox proportional hazards model; Hazard Ratio (HR) = 1.271, 95% CI 2-sided [0.573 to 2.819]

8. Secondary Outcome: Blood Glucose Levels for Patients Reporting Severe Hypoglycemia at Months 6, 12 and 18
Description: A severe hypoglycemic event was defined as an event with 1 of the following symptoms: "memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL or prompt recovery after oral carbohydrate, i.e. glucose, or glucagon administration. Summary statistics of blood glucose level (mg/dL) are provided by treatment group at each time point for patients reporting severe hypoglycemia.
Time Frame: Months 6 (week 26±2), 12 (week 52±2) and 18 (week 78±2)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 18 | 7
mg/dL
  Month 6 | 48.11 (4.73) | 51.00 (3.94)
  Month 12 | 48.71 (4.75) | 49.57 (5.71)
  Month 18 | 48.27 (4.90) | 50.13 (5.51)

9. Secondary Outcome: Change From Baseline in Average (Previous 3 Days) Daily Insulin Requirements (IU/kg/Day) at Months 6,12 and 18
Description: For the purpose of this study, daily insulin is averaged over the previous 3 days.Insulin requirement (IU/kg/day averaged over the previous 3 days) was to be recorded to Months 6, 12 and 18.
  Patients were admitted to intensive diabetes management, according to current ADA recommendation [2014]. Patients were instructed to self-monitor their glucose values at least 4 times a day and to report (glucose meter/log) outcome to the diabetes management team. Insulin intake was adjusted to target HbA1c levels of less than 7% and self-monitored (fingerstick):
  * pre-prandial blood glucose of 70-130 mg/dL
  * post-prandial blood glucose < 180 mg/dL
  * bed-time blood glucose of 110-150 mg/dL
Time Frame: Months 6 (26±2 weeks), 12 (52±2 weeks) and 18 (78±2 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 16 | 7
IU/kg/day
  Month 6: number analyzed (Participants) | 16 | 6
  Month 6 | -0.209 (0.644) | -0.028 (0.228)
  Month 12: number analyzed (Participants) | 15 | 7
  Month 12 | -0.183 (0.661) | 0.024 (0.271)
  Month 18: number analyzed (Participants) | 15 | 7
  Month 18 | -0.183 (0.639) | -0.005 (0.342)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6 for change from baseline; Test type: Superiority; p = 0.320, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 12 for change from baseline; Test type: Superiority; p = 0.398, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Comparison at month 18 for change from baseline; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

10. Secondary Outcome: Change From Baseline in Estimated Glucose Disposal Rate (eGDR) at Months 6, 12 and 18
Description: Estimated Glucose Disposal Rate (eGDR) is a marker for the Assessment of Insulin Resistance and a validated clinical tool for estimating insulin sensitivity in type 1 diabetes.
Time Frame: Months 6 (26±2 weeks), 12 (52±2 weeks) and 18 (78±2 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 15 | 7
mg/kg/min
  Month 6 | 0.418 (0.815) | 0.367 (0.816)
  Month 12: number analyzed (Participants) | 14 | 6
  Month 12 | 0.067 (1.504) | 0.623 (0.862)
  Month 18: number analyzed (Participants) | 15 | 6
  Month 18 | 0.242 (1.142) | -0.238 (1.255)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Comparison at month 6 for change from baseline; Test type: Superiority; p = 0.892, t-test, 2 sided — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Comparison at month 12 for change from baseline; Test type: Superiority; p = 0.412, t-test, 2 sided — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Comparison at month 18 for change from baseline; Test type: Superiority; p = 0.371, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

11. Secondary Outcome: Number of Patients With at Least One Adverse Events (AEs), Serious or Not Serious
Description: An AE is any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the trial intervention.
  A serious adverse event is an adverse event that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect.
Time Frame: Throughout the study up to 18 months
Population: SAF population: The Safety (SAF) population consisted of all randomized patients who received at least one dose of the IMP. The SAF population was analyzed according to the actual treatment received and was used to present results on safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 18 | 7
Participants
  any TEAE | 12 | 5
  serious TEAE | 1 | 0
  non-serious TEAE | 12 | 5
  TEAEs leading to IMP discontinuation | 1 | 1
  TEAEs leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study, from the baseline to the study termination (from cycle 1 up to Month 12) and follow-up (Month 18)
Arm/Group | Ladarixin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/7
Other Adverse Events (participants affected / at risk) | 12/18 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladarixin (N=18) | Placebo (N=7)
primary hyperparathyroidism (Endocrine disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladarixin (N=18) | Placebo (N=7)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (5) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasal herpes (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (8) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorders (Nervous system disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Normocytic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Occult blood (Investigations) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Amenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Fixed eruption (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The enrolment was stopped on March,28, 2022 due to low enrolment rate at the randomization of the 25th patient. Due to the trial early termination, efficacy analyses were reduced given the limited sample size of the study vs with the one expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT04899271/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT04899271/SAP_001.pdf